CLINICAL TRIAL: NCT02203877
Title: Nutritional Intervention Study, Randomized, Double-blind, Parallel Group to Evaluate the Effect of Lactobacillus Fermentum CECT5716 Consumption on the Incidence of Mastitis
Brief Title: Evaluation of Lactobacillus Fermentum CECT5716 on the Incidence of Mastitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P032
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2014-07

CONDITIONS: Mastitis
MeSH Terms: conditions — Mastitis | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Placebo Comparator): 1 capsule/day for 16 weeks
  Interventions: Dietary Supplement: Maltodextrin
- Lactobacillus fermentum CECT5716 (Experimental): L.fermentum 3,00E+09cfu/day. 1 capsule/day for 16 weeks
  Interventions: Dietary Supplement: Lactobacillus fermentum CECT5716

INTERVENTIONS:
Dietary Supplement: Lactobacillus fermentum CECT5716 — Intervention with a probiotic strain in form of a daily capsule containing 3x109cfu/capsule.
  Arms: Lactobacillus fermentum CECT5716
Dietary Supplement: Maltodextrin — Intervention with a daily capsule containing maltodextrin as placebo
  Arms: Maltodextrin

SUMMARY:
To evaluate the effect of the consumption of Lactobacillus fermentum CECT5716 on mastitis incidence.

DETAILED DESCRIPTION:
Previous studies have demonstrated that L. fermentum CECT5716, a probiotic strain previously isolated from breast milk, can be used as an effective treatment of mastitis and painful breastfeeding by reducing pathogen counts in breast milk. This is a randomized double blinded controlled study to evaluate the effect of L.fermentum CECT5716 on mastitis incidence and Staphylococcus load in breast milk. Women will be recruited 1-6 days after child birth and distributed into two groups: Probiotic group receiving 1 capsule/day containing L.fermentum 3x109cfu; Control group receiving 1 placebo capsule/day containing maltodextrin. The intervention period is 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between 18 and 40 years with development of normal pregnancy Birth between 37 and 42 weeks of gestation. Women who have received antibiotic treatment between 48 hours before and 48 hours after childbirth (one dose is sufficient for inclusion regardless of the type of antibiotic).

Childbirth took place 1-7 days prior to recruitment.. With firm intention to breast-feed their children for at least 16 weeks..

Exclusion Criteria:

* - Mammary pathologies that hinder or preclude breastfeeding.
* Low expectation of adherence to the study protocol.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 625 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
incidence of mastitis | up to 16 weeks
  mastitis was defined as at least two out of the three breast symptoms (pain, redness, lump) and at least one of fever or flu-like symptoms (shivering, hot sweats or aches)

SECONDARY OUTCOMES:
evaluation of breast pain | at times 0, 4, 8, 12 and 16 weeks
  For pain evaluation a score from 1 (no pain) to 10 (extremely pain)

OTHER OUTCOMES:
microbiota breast milk | at time 0 and 16 weeks
  DNA will be extracted from breast milk samples. Staphylococcus genus, Streptococcus and Lactobacillus will be evaluated by qPCR with specific probes designed to quantify these bacterial genus.
fecal microbiota of infants | at 0 and 16 weeks
  DNA will be extracted from infant´s feces samples. Lactobacillus, bifidobacterium, clostridium, bacteroides will be evaluated by qPCR with specific probes designed to quantify these bacterial genus.
growth of infants | at 0 and 16 weeeks
  Weight, length and head circumference will be measured in infants at the beginning and at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juristo Fonollá, PhD, Study Chair — Biosearch S.A.
Locations (1):
- Hospital Virgen de las Nieves, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crepinsek MA, Taylor EA, Michener K, Stewart F. Interventions for preventing mastitis after childbirth. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD007239. doi: 10.1002/14651858.CD007239.pub4. PMID 32987448
- [Derived] Pastor-Villaescusa B, Hurtado JA, Gil-Campos M, Uberos J, Maldonado-Lobon JA, Diaz-Ropero MP, Banuelos O, Fonolla J, Olivares M; PROLAC Group. Effects of Lactobacillus fermentum CECT5716 Lc40 on infant growth and health: a randomised clinical trial in nursing women. Benef Microbes. 2020 May 11;11(3):235-244. doi: 10.3920/BM2019.0180. Epub 2020 Mar 27. PMID 32216468